CLINICAL TRIAL: NCT03850561
Title: The Effect of Two Doses of Coenzyme Q10 on Seminal Fluid Parameters and Antioxidant Status: A Randomised Controlled Trial
Brief Title: Effect of Two Doses of Coenzyme Q10 on Seminal Fluid and Semen Antioxidant Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sumer (Other)
Responsible Party: Principal Investigator, Dr. Ahmed T Alahmar, Principal Investigator, University of Sumer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2018/8878
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Male Infertility
Keywords: Male infertility; Coenzyme Q10; Antioxidants
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q10 200 (Active Comparator): Coenzyme Q10 200mg/day for 3 months
  Interventions: Dietary Supplement: Coenzyme Q10 200
- Coenzyme Q10 400 (Active Comparator): Coenzyme Q10 400mg/day for 3 months
  Interventions: Dietary Supplement: Coenzyme Q10 400

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 200 — Coenzyme Q10 200 mg/day
  Arms: Coenzyme Q10 200
Dietary Supplement: Coenzyme Q10 400 — Coenzyme Q10 400 mg/day
  Arms: Coenzyme Q10 400

SUMMARY:
The study was conducted to assess the impact of two doses of coenzyme Q10 on seminal fluid parameters and antioxidant status in infertile men.

DETAILED DESCRIPTION:
The aim of this study was to assess the impact of two doses of coenzyme Q10 on seminal fluid parameters and antioxidant status in infertile men with idiopathic oligoasthenoteratospermia.

ELIGIBILITY:
Inclusion Criteria:

* History of infertility of at least 12 months despite regular unprotected intercourse.

Oligoasthenoteratospermia was diagnosed by semen analysis showing abnormal sperm concentration (<15 million/ml), progressive motility (<32%), total motility (<40%) and morphology (<30% WHO criteria) as defined by WHO manual for semen analysis 2010

Exclusion Criteria:

* Azoospermia,
* Varicocele,
* Genital tract infection,
* Cryptorchidism,
* Testicular trauma or scrotal surgery,
* Endocrine disorder,
* Systemic illness,
* Smoking
* The presence of female factor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male Infertility
Enrollment: 65 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Semen volume (WHO 2010 guidelines) | 3 months
  Semen volume in ml
Sperm concentration in semen (WHO 2010 guidelines) | 3 months
  Sperm concentration in million/ml
Sperm motility in semen (WHO 2010 guidelines) | 3 months
  Sperm motility (%)
Sperm morphology in semen (WHO 2010 guidelines) | 3 months
  Normal sperm morphology (%)
Seminal plasma TAC | 3 months
  Seminal plasma total antioxidant capacity in mmol/ml
Seminal plasma CAT | 3 months
  Seminal plasma catalase in U/ml
Seminal plasma SOD | 3 months
  Superoxide dismutase in U/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T Alahmar, MBChB, MSC, Principal Investigator — University of Sumer, Iraq
Locations (1):
- Fertility Unit, Babyl, Hillah, Iraq

IPD SHARING:
Plan to Share IPD: No
Patients data are anonymous and in hold with the principal investigator

REFERENCES:
- [Background] Alahmar AT. The effects of oral antioxidants on the semen of men with idiopathic oligoasthenoteratozoospermia. Clin Exp Reprod Med. 2018 Jun;45(2):57-66. doi: 10.5653/cerm.2018.45.2.57. Epub 2018 Jun 29. PMID 29984205
- [Background] Alshahrani S, Aldossari K, Al-Zahrani J, Gabr AH, Henkel R, Ahmad G. Interpretation of semen analysis using WHO 1999 and WHO 2010 reference values: Abnormal becoming normal. Andrologia. 2018 Mar;50(2). doi: 10.1111/and.12838. Epub 2017 Aug 3. PMID 28771785
- [Background] Nadjarzadeh A, Shidfar F, Amirjannati N, Vafa MR, Motevalian SA, Gohari MR, Nazeri Kakhki SA, Akhondi MM, Sadeghi MR. Effect of Coenzyme Q10 supplementation on antioxidant enzymes activity and oxidative stress of seminal plasma: a double-blind randomised clinical trial. Andrologia. 2014 Mar;46(2):177-83. doi: 10.1111/and.12062. Epub 2013 Jan 7. PMID 23289958